CLINICAL TRIAL: NCT05670665
Title: Impact of Threatened Preterm Labour in Fetal Cardiovascular and Metabolic Programming
Brief Title: Impact of Threatened Preterm Labour in Fetal Cardiovascular and Metabolic Programming (SHs)
Acronym: SHs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Cristina Paules, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Other Study IDs: Superhearts Study
Record Dates: First submitted 2022-11-03; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Obstetric Labor, Premature
Keywords: Threatened preterm labor; Prematurity; Cardiac remodelling; Cardiac function
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood from umbilical cord
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-exposed: Low-risk, singleton pregnancies.
- Exposed: Singleton pregnancies that are admitted to hospital due to threatened preterm labor or preterm premature rupture of membranes.
  Interventions: Other: Threatened preterm labor

INTERVENTIONS:
Other: Threatened preterm labor — Presence of uterine contractions and cervical shortening between 24+0 and 36+6 weeks of gestation and/or rupture of the membranes between 24+0 and 36+6 weeks of gestation.
  Groups: Exposed

SUMMARY:
The goal of this observational study is to learn about cardiac function and remodelling and metabolomic profiles in fetuses and infants who were exposed to a threatened preterm labor (TPL) during pregnancy.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* Evaluate the impact of threated preterm labour in cardiovascular and metabolic programming in fetal life and early infancy.
* Describe prenatal and postnatal patterns of cardiac remodelling associated to threatened preterm labour.
* Describe fetal growth patterns associated to threatened preterm labour.
* Describe metabolomic profiles in umbilical cord blood associated to cardiovascular programming in fetuses exposed to threatened preterm labour.

The study's main tasks are:

* To perform an antenatal echocardiography of the exposed cohort is performed during the admission due to TPL or preterm spontaneous rupture of membranes (SRM).
* All participants are asked to fill a diet and stress questionnaire.
* To collect cord blood at the time of delivery.
* To perform a postnatal echocardiography six months after birth.

Researchers will compare fetuses and infants who were exposed to TPL to those who were not exposed to TPL during pregnancy to see if threre are any differences in cardiac function and remodelling.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies.
* Study patients must be 18 years or older
* Good understanding of Spanish

Exclusion Criteria:

* Multiple pregnancies
* Major fetal defects or anomalies
* Underlying process that can cause a preterm labour
* Iatrogenic preterm labour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are elegible for this study
Study Population: Exposed cohort: women older than 18 years-old who have a singleton pregnancy and who are admitted to our unit due to TPL or preterm SRM are offered to participate in the study. Non-exposed cohort: women older than 18 years-old who have a singleton pregnancy and who attend our low-risk antenatal clinic are selected randomly and offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fetal cardiac sphericity index | 24 - 36+6 weeks of gestation
  2-D mode
Fetal cardiac diameters | 24 - 36+6 weeks of gestation
  Measurement of atrial and ventricular longitudinal and transverse diameters with 2-D mode
Fetal ventricular and atrial areas | 24 - 36+6 weeks of gestation
  2-D mode
Fetal cardiac ejection fraction | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal cardiac ejection volume | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal cardiac filling and ejection time fractions | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal cardiac debit | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal mitral and tricuspid annular plane systolic excursion (MAPSE and TAPSE) | 24 - 36+6 weeks of gestation
  M-mode
Fetal cardiac E/A ratios | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal cardiac isovolumetric relaxation time | 24 - 36+6 weeks of gestation
  Pulsed-Doppler
Fetal Doppler | 24 - 36+6 weeks of gestation
  Measurement of umbilical artery pulsatility index (PI), medial cerebral artery PI and systolic peak (SP), ductus venosus PI, and mean uterine arteries PI using pulsed-Doppler
Fetal growth | 24 - 36+6 weeks of gestation
  Hadlock formula
ProBNP, troponin and cystatin levels in cord blood | Third stage of labor
  Electrochemiluminescence immunoassay
Estimated left ventricular myocardial mass | 6 months
  2D echochardiography
Left ventricular muscle index | 6 months
  2D echochardiography
Left ventricular end-diastolic volume | 6 months
  2D echochardiography
Left ventricular ejection fraction | 6 months
  2D echochardiography
Infant global cardiac longitudinal strain rate | 6 months
  Using echocardiography in order to measure myocardial function
Infant cardiac strain rate imaging | 6 months
  Using echocardiography in order to measure myocardial function

SECONDARY OUTCOMES:
Adherence to Mediterranean diet | 24 - 36+6 weeks of gestation
  Validated 14-item PREDIMED (Prevención con dieta mediterránea) questionnaire. Minimum value is 0. Maximum value is 14. We expect a better outcome the higher the score.
Maternal stress levels | 24 - 36+6 weeks of gestation
  Perceived Stress Scale (PSS). Minimum score: 0. Maximum score: 40. We expect to find worse outcomes with higher scores.
Maternal anxiety levels | 24 - 36+6 weeks of gestation
  State-Trait Anxiety Index (STAI). Minimum score: 20. Maximum score: 80. We expecto to find worse outcomes with higher scores.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Paules, Principal Investigator — IIS Aragon, Hospital Clinico Universitario Lozano Blesa
Locations (1):
- Hospital Clinico Universitario Lozano Blesa, Zaragoza, Spain

REFERENCES:
- [Derived] Abadia-Cuchi N, Clavero-Adell M, Gonzalez J, Medel-Martinez A, Fabre M, Ayerza-Casas A, Youssef L, Lerma-Irureta J, Maestro-Quibus P, Rodriguez-Calvo J, Ruiz-Martinez S, Lerma D, Schoolermer J, Oros D, Paules C. Impact of suspected preterm labour in foetal cardiovascular and metabolic programming: a prospective cohort study protocol. BMJ Open. 2024 Nov 24;14(11):e087430. doi: 10.1136/bmjopen-2024-087430. PMID 39581725